CLINICAL TRIAL: NCT03158168
Title: Intralesional Candidal Antigen Versus Intralesional Zinc Sulphate in Treatment of Cutaneous Warts, A Randomized Clinical Trial
Brief Title: Intralesional Candidal Antigen Versus Intralesional Zinc Sulphate in Treatment of Cutaneous Warts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAAbdelsalam, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: candida and zinc in warts
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — PRA1 protein, Candida albicans; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The first group will receive Intralesional injection of Candidal antigen with a dose of (0.1ml -0.3ml) by insulin syringe in the largest wart at the first visit.( Only those patients who showed a positive response to the Candida test antigen).I njections will be repeated for all patients into the same lesion every 3 weeks for three treatment sessions. Follow up for next six months for any recurrences.
  Storage: A 1ml multidose vial of candidal antigen (Candin) which is an intradermal test antigen, stored between 2c-8c.
  Interventions: Drug: Candida Antigen
- control group (Active Comparator): The second group will receive an IL injection of 2%Zn sulfate with a dose of (0.1ml-0.3ml) by insulin syringe ,in the largest one .the wart is injected with the solution till blanching or bleb formation. Subcutaneous injections and acral parts such as fingers and toes will be avoided, as it may cause vascular necrosis [19]. Injections will be repeated for all patients into the same lesion every 2 weeks for three treatment sessions.Follow up for next six months for any recurrences.
  Preparation of 2% zinc sulfate: A measure of 2g. of zinc sulfate powder is to be dissolved in 100 ml of sterile distilled water and autoclaved at 95c for 20 min(20).
  Interventions: Drug: Zinc Sulfate

INTERVENTIONS:
Drug: Candida Antigen — Candida Albicans Antigen injection
  Arms: study group
Drug: Zinc Sulfate — Zinc Sulfate injection
  Arms: control group

SUMMARY:
Warts are common and infectious viral diseases of the skin and are prevalent worldwide. Warts are caused by the human papilloma virus (HPV), which has more than 100 strains; some of them are known to be premalignant .Although warts can appear at any age, they are more common in children and adolescents. The prognosis of warts cannot be predicted. In some patients they may spontaneously disappear, whereas others show persistence and progression with spreading to other body sites, leading to physical and emotional distress to the patients. [ 1 ].

DETAILED DESCRIPTION:
Forty percent of children spontaneously clear in two years without treatment owing to natural immunity [ 2,3.]. However, warts can persist and increase in size and number [2] .

Warts may reflect a localized or systemic cell-mediated immune (CMI) deficiency to HPV. Various reasons like lack of production of memory T cells to target HPV infection, failure of clonal expansion of lymphocytes to adequate stimulation, inability of T lymphocytes to traffic to sites of infection and weak effector response mechanism have been hypothesized. [4] .] Consequently, warts are particularly exuberant in patients with Hodgkin's disease, AIDS and those on immunosuppressant [ 5 ].

The conventional modalities in treatment of warts include destructive therapies such as salicylic acid, trichloroacetic acid, cryotherapy, silver nitrate, phenol, canthiridin, electrocautary, surgical interventions and lasers; antiproliferative agents such as bleomycin, vitamin D analogs, podophyllin, and 5-fluro uracil; antiviral agents such as cidofovir and retinoids. Because of the cumbersome nature of these procedures and a high risk of recurrence, immunotherapy is becoming more and more popular, especially in the treatment of refractory cutaneous and genital warts [ 6 ] . It enhances recognition of the virus by the immune system. This allows not only clearing of the treated wart, and frequently warts at distant anatomic sites, but also may prevent future clinical infection [ 7 ] .

Immunotherapy in warts can be administered by various methods. The first method is topical application of certain inorganic molecules that are capable of eliciting a contact hypersensitivity reaction with secondary activation of an immunological response [ 8 ] . A second modality is the use of oral immune modulators such as cimetidine and zinc(10mg/kg/day for 2months) [ 9 , 10 ] .

A third method is Intralesional injection of immunotherapeutic agent that utilizes the ability of the immune system to mount a delayed type hypersensitivity response to various antigens and also the wart tissue leading to production of Th1 cytokines which activate cytotoxic and natural killer cells to eradicate HPV infection. This clears not only the local warts but also distant warts unlike traditional wart therapies [ 11 ] .

There are a few side effects reported by most of the studies. The most common side effect was pain and discomfort during injection, however, serious side effects such as vitiligo-like depigmentation and painful purple digit have also been reported [ 12 ] .

Zinc is important for immune regulation as it stimulates the leucocytes and natural killer cells. It has been shown that there is a deficiency of zinc in patients with multiple or recurrent warts [ 13 ,14 ].The use of zinc in treatment of warts was proven in many studies either in the topical form or systemic oral therapy [ 15 ].. However, Little studies have utilized intralesional injection of 2% zinc sulfate solution for the treatment of common wart one of them was of [16] .

ELIGIBILITY:
Inclusion Criteria:- patients with ages ranging from 10 to 40 years with cutaneous common or planter wart ,

* or were either resistant to treatment
* or had relapsed at least once after treatment with any of the tissue-destructive modalities

Exclusion Criteria:.- Patients with any evidence of immunosuppressant,

* eczematous skin disorder,
* those with any history of hypersensitivity to Candida albicans antigen,
* pregnant or lactating women,
* and those who received any wart treatment 1 month before the start of the study will be excluded from the study

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
complete resolution of the injected wart | 9 weeks
  by photography

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch MD, Cliffe J, Morris-Jones R. Management of cutaneous viral warts. BMJ. 2014 May 27;348:g3339. doi: 10.1136/bmj.g3339. No abstract available. PMID 24865780
- [Background] Bacelieri R, Johnson SM. Cutaneous warts: an evidence-based approach to therapy. Am Fam Physician. 2005 Aug 15;72(4):647-52. PMID 16127954
- [Background] Gibbs S, Harvey I. Topical treatments for cutaneous warts. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD001781. doi: 10.1002/14651858.CD001781.pub2. PMID 16855978
- [Background] Scheinfeld N. Treatment of molluscum contagiosum: a brief review and discussion of a case successfully treated with adapelene. Dermatol Online J. 2007 Jul 13;13(3):15. PMID 18328209
- [Background] Sinha S, Relhan V, Garg VK. Immunomodulators in warts: Unexplored or ineffective? Indian J Dermatol. 2015 Mar-Apr;60(2):118-29. doi: 10.4103/0019-5154.152502. PMID 25814698
- [Background] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231
- [Background] Johnson SM, Roberson PK, Horn TD. Intralesional injection of mumps or Candida skin test antigens: a novel immunotherapy for warts. Arch Dermatol. 2001 Apr;137(4):451-5. PMID 11295925
- [Background] Silverberg NB, Lim JK, Paller AS, Mancini AJ. Squaric acid immunotherapy for warts in children. J Am Acad Dermatol. 2000 May;42(5 Pt 1):803-8. doi: 10.1067/mjd.2000.103631. PMID 10775858
- [Background] Rogers CJ, Gibney MD, Siegfried EC, Harrison BR, Glaser DA. Cimetidine therapy for recalcitrant warts in adults: is it any better than placebo? J Am Acad Dermatol. 1999 Jul;41(1):123-7. doi: 10.1016/s0190-9622(99)70421-4. PMID 10411426
- [Background] Orlow SJ, Paller A. Cimetidine therapy for multiple viral warts in children. J Am Acad Dermatol. 1993 May;28(5 Pt 1):794-6. doi: 10.1016/s0190-9622(09)80278-8. No abstract available. PMID 8496433
- [Background] Nofal A, Nofal E. Intralesional immunotherapy of common warts: successful treatment with mumps, measles and rubella vaccine. J Eur Acad Dermatol Venereol. 2010 Oct;24(10):1166-70. doi: 10.1111/j.1468-3083.2010.03611.x. PMID 20202055
- [Background] Perman M, Sterling JB, Gaspari A. The painful purple digit: an alarming complication of Candida albicans antigen treatment of recalcitrant warts. Dermatitis. 2005 Mar;16(1):38-40. PMID 15996350
- [Background] Raza N, Khan DA. Zinc deficiency in patients with persistent viral warts. J Coll Physicians Surg Pak. 2010 Feb;20(2):83-6. PMID 20378032
- [Background] Lopez-Garcia DR, Gomez-Flores M, Arce-Mendoza AY, de la Fuente-Garcia A, Ocampo-Candiani J. Oral zinc sulfate for unresponsive cutaneous viral warts: too good to be true? A double-blind, randomized, placebo-controlled trial. Clin Exp Dermatol. 2009 Dec;34(8):e984-5. doi: 10.1111/j.1365-2230.2009.03623.x. No abstract available. PMID 20055878
- [Derived] Youssef EMK, Eissa MAA, Bakr RM. Intralesional Candida albicans antigen versus intralesional zinc sulfate in treatment of cutaneous warts. Arch Dermatol Res. 2023 Jul;315(5):1305-1314. doi: 10.1007/s00403-022-02499-w. Epub 2022 Dec 26. PMID 36567351